CLINICAL TRIAL: NCT05755399
Title: Feasibility of Transcranial Focused Ultrasound to Measure Brain Tumor
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: Feasibility
Record Dates: First submitted 2023-01-16; First posted 2023-03-06 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-09

CONDITIONS: Cranial Neurosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Experimental group (Experimental): Participants scheduled for brain surgery
  Interventions: Device: Brain imaging using transcranial focused ultrasound (tFUS)

INTERVENTIONS:
Device: Brain imaging using transcranial focused ultrasound (tFUS) — All enrolled patients will be imaged using the MRI as standard of care. The patient will additionally be imaged using the tFUS system, ICC HIFU Synthesizer. Total imaging time will be limited to 15 minutes. Following image acquisition by the ultrasound, the standard of care surgery will be performed.

SUMMARY:
Transcranial focused ultrasound (tFUS) offers a platform for non-invasive imaging and treatment of the brain and pathology of the brain -- allowing high resolution imaging in both spatial and temporal dimensions. Compared with the gold- standard for brain imaging, magnetic resonance imaging (MRI), ultrasound offers reduced contrast while providing improved sampling in time through a significantly more cost-effective approach. In addition, while MRI is used to guide invasive treatments, only ultrasound can offer treatments through three primary mechanisms: 1) neuromodulation, 2) blood brain barrier modulation, and thermal/mechanical ablation through high intensity focused ultrasound (HIFU). All three treatment options require targeting therapy through the skull, which remains a barrier to clinical translation. This proposal is to test the feasibility of acquiring noninvasive targeting imaging intraoperatively prior to clinically indicated cranial neurosurgery. By acquiring volumetric ultrasound images while coregistered to previously obtained stereotactic magnetic resonance imaging, the study will be able to compare the ability of tFUS to identify and focus on brain pathology.

ELIGIBILITY:
Inclusion Criteria:

* Able to undergo informed consent
* Scheduled and present for brain surgery
* General Anesthesia planned
* Neuronavigation used for surgery
* Thin cut post-contrast imaging available for coregistration
* At least 18 years of age

Exclusion Criteria:

* Awake craniotomy planned
* Unhealed wounds or infection of scalp
* Diseases and conditions that would increase the morbidity and mortality of craniotomy and tumor resection (e.g. cardiopulmonary issues) in the opinion of the PI.
* Pregnancy (also generally required for surgery)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2023-10-19 (Actual); Primary Completion 2026-05-01 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Test feasibility | baseline
  For each participant feasibility is defined as 1 when any ultrasound slices are obtained and segmented. If tumor segmentation cannot be performed then this will be reported as 0, meaning not feasible. The result at the group level is a feasibility measure, i.e., the proportion of participants for whom the protocol was feasible.

SECONDARY OUTCOMES:
Volume assessment | Baseline
  three-dimensional reconstructions of MRI slices will be manually segmented, resulting in a tumor volume that will be compared with MRI-segmented tumor volume.
Morphology assessment | Baseline
  three-dimensional ultrasound and MRI reconstructions will be co-registered onto a three dimensional grid and compared. The ratio of the MRI and FUS derived volumes will be computed, resulting in a distribution. A value of one for this ratio indicates perfect agreement.

CONTACTS AND LOCATIONS:
Overall Officials: David Darrow, MD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No